CLINICAL TRIAL: NCT03751553
Title: Obstetrical Gel and Its Impact in Shortening the Duration of Labor in Women Undergoing a Vaginal Birth After Cesarean (VBAC):a Randomized Controlled Trial
Brief Title: Obstetrical Gel and Its Impact in Shortening the Duration of Labor in Women Undergoing a Vaginal Birth After Cesarean (VBAC)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: obstetrical gel
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Duration of Labor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obstetric gel group (Experimental): they will have the standard care during labor and delivery with the vaginal application of the obstetrical gel.
  Interventions: Drug: obsteric gel(k-Y jelly)
- no intervention group (No Intervention): they will receive the standard care during labor and delivery without the use of the obstetrical gel

INTERVENTIONS:
Drug: obsteric gel(k-Y jelly) — A sterile obstetric gel( K-Y Jelly 82GM; manufactured by Johnson& Johnson) will be used for this trial. The obstetric gel is a birth gel with no pharmacologic effects that have purely physical activity. Starting with the first vaginal examination the obstetric gel will be used. After each vaginal examination, 3-5 mL of obstetric gel will be introduced into the vaginal birth canal in the area in front of the child manually or using the sterile obstetric gel applicator without any manipulation or massage.
  Arms: obstetric gel group

SUMMARY:
The objective of our study is to investigate whether the use of obstetric gel shortens the first and second stage of labor and exerts a protective effect on the lower genital tract in women undergoing a Vaginal Birth After Cesarean (VBAC).

DETAILED DESCRIPTION:
Recent literature shows that birth injury is associated with postpartum pelvic floor dysfunction (pelvic organ prolapse and fecal and urinary incontinence). Prolonged labor, namely during the 2nd stage, is one of the main obstetric risk factors responsible for anal sphincter rupture and fecal incontinence. In addition, it is associated with increased maternal and neonatal morbidities including increased risk of lower genital tract lacerations. In an effort to shorten labor and decrease lower genital tract trauma many techniques have been investigated.

ELIGIBILITY:
Inclusion Criteria:

* • Age between 18 and 40 years

  * Women who have had only one prior cesarean birth with no previous vaginal delivery, are eligible for VBAC and plan to attempt a VBAC after counseling.
  * Singleton baby in vertex presentation
  * Low-risk pregnancy at term (37-41 weeks of gestation)
  * Estimated birth weight between 2000 g and 4500 g (clinically or by sonography)
  * Signed written informed consent

Exclusion Criteria:

* • Contraindications for vaginal delivery (placenta previa, active herpes infection, etc…)

  * Suspected amniotic infection (fever, foul-smelling discharge, fetal tachycardia, abdominal pain)
  * A non-reassuring fetal heart tracing
  * Prolonged rupture of the membranes (24 hours)
  * Suspected major fetal malformations
  * Suspected cephalopelvic disproportion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2018-12-30 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
length of the second stage of labor | 1 hour
  the length of the second stage of labor starting from full cervical dilatation till delivery of the fetus will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University
Locations (1):
- Ahmed Ashour, Giza, Egypt